CLINICAL TRIAL: NCT00134264
Title: Phase 3 Multi Center, Double Blind, Randomized, Parallel Group Evaluation Of The Fixed Combination Torcetrapib/Atorvastatin, Administered Orally, Once Daily (Qd), Compared With Atorvastatin Alone, On The Occurrence Of Major Cardiovascular Events In Subjects With Coronary Heart Disease Or Risk Equivalents
Brief Title: A Study Examining Torcetrapib/Atorvastatin And Atorvastatin Effects On Clinical CV Events In Patients With Heart Disease
Acronym: ILLUMINATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091043
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-01

CONDITIONS: Coronary Disease; Diabetes Mellitus
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To demonstrate if torcetrapib/atorvastatin can reduce the risk for major cardiovascular disease events, when compared to atorvastatin alone, in patients with coronary heart disease or risk equivalents

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of coronary heart disease or risk equivalents that place the patient at high risk for cardiovascular disease events

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluationof response, or render unlikely that the subject would complete the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15067 (Actual)
Dates: Start 2004-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
The time to first occurrence of a major cardiovascular disease event

SECONDARY OUTCOMES:
Various composites of major cardiovascular disease events and other lipid parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (221):
- United States (95):
  - Pfizer Investigational Site, Alabaster, Alabama
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Gilbert, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Modesto, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Rosa, California
  - Pfizer Investigational Site, Tustin, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Longmont, Colorado
  - Pfizer Investigational Site, Guilford, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Coral Gables, Florida
  - Pfizer Investigational Site, Fort Meyers, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Jacksonville Beach, Florida
  - Pfizer Investigational Site, Lakeland, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Pensacola, Florida
  - Pfizer Investigational Site, Port Charlotte, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, West Palm Beach, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Aurora, Illinois
  - Pfizer Investigational Site, Blue Island, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Fort Wayne, Indiana
  - Pfizer Investigational Site, Davenport, Iowa
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Witchita, Kansas
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Covington, Louisiana
  - Pfizer Investigational Site, Marrero, Louisiana
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bel Air, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Westminster, Maryland
  - Pfizer Investigational Site, Abington, Massachusetts
  - Pfizer Investigational Site, Haverhill, Massachusetts
  - Pfizer Investigational Site, Natick, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Paul, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Papillon, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Concord, New Hampshire
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Manchester, New Hampshire
  - Pfizer Investigational Site, Elmer, New Jersey
  - Pfizer Investigational Site, Haddon Heights, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Mansfield, Ohio
  - Pfizer Investigational Site, Sandusky, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Beaver, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Beaumont, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Plano, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Burien, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Australia (25):
  - Pfizer Investigational Site, Concord, New South Wales
  - Pfizer Investigational Site, East Gosford, New South Wales
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Wollongong, New South Wales
  - Pfizer Investigational Site, Chermside, Queensland
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Woolloongabba, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Bedford Park, South Australia
  - Pfizer Investigational Site, Woodville, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Fitzroy, Victoria
  - Pfizer Investigational Site, Footscray, Victoria
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Prahran, Victoria
  - Pfizer Investigational Site, Fremantle, Western Australia
  - Pfizer Investigational Site, Joondalup, Western Australia
  - Pfizer Investigational Site, Camperdown
  - Pfizer Investigational Site, Darlinghurst
  - Pfizer Investigational Site, Geelong
  - Pfizer Investigational Site, Launceston, Tas
  - Pfizer Investigational Site, Melbourne
  - Pfizer Investigational Site, Nedlands
  - Pfizer Investigational Site, Perth
  - Pfizer Investigational Site, Southport
- Canada (16):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Vancouver, British Columbia
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Halifax, Nova Scotia
  - Pfizer Investigational Site, Cornwall, Ontario
  - Pfizer Investigational Site, Newmarket, Ontario
  - Pfizer Investigational Site, Oshawa, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Scarborough Village, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Sainte-Foy, Quebec
  - Pfizer Investigational Site, Sherbrooke, Quebec
  - Pfizer Investigational Site, Ste-foy, Quebec
  - Pfizer Investigational Site, St. John's
- Netherlands (23):
  - Pfizer Investigational Site, 's-Hertogenbosch
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, AN Rotterdam
  - Pfizer Investigational Site, Apeldoorn
  - Pfizer Investigational Site, Arnhem
  - Pfizer Investigational Site, Breda
  - Pfizer Investigational Site, Cappelle Aan Den IJssel
  - Pfizer Investigational Site, Delft
  - Pfizer Investigational Site, Eindhoven
  - Pfizer Investigational Site, Goes
  - Pfizer Investigational Site, Gouda
  - Pfizer Investigational Site, Groningen
  - Pfizer Investigational Site, Heerlen
  - Pfizer Investigational Site, Hoorn
  - Pfizer Investigational Site, Leiden
  - Pfizer Investigational Site, Maastricht
  - Pfizer Investigational Site, Nijmegen
  - Pfizer Investigational Site, Rotterdam
  - Pfizer Investigational Site, Sittard
  - Pfizer Investigational Site, Utrecht
  - Pfizer Investigational Site, Velp
  - Pfizer Investigational Site, Venlo
  - Pfizer Investigational Site, Zoetermeer
- Spain (18):
  - Pfizer Investigational Site, Almería, Almeria
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Sant Coloma de Gramenet, Barcelona
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Jerez de la Frontera, Cadiz
  - Pfizer Investigational Site, Santander, Cantabria
  - Pfizer Investigational Site, Ciudad Real, Ciudad Real
  - Pfizer Investigational Site, Granada, Granada
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Ferrol, La Coruna
  - Pfizer Investigational Site, Santiago de Compostela, La Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Málaga, Malaga
  - Pfizer Investigational Site, Seville, Sevilla
  - Pfizer Investigational Site, Valencia, Valencia
  - Pfizer Investigational Site, Zaragoza, Zaragoza
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Salamanca
- Sweden (20):
  - Pfizer Investigational Site, Borås
  - Pfizer Investigational Site, Eskilstuna
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Hässleholm
  - Pfizer Investigational Site, Helsingborg
  - Pfizer Investigational Site, Karlshamn
  - Pfizer Investigational Site, Köping
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Luleå
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Mölndal
  - Pfizer Investigational Site, Norrköping
  - Pfizer Investigational Site, Östersund
  - Pfizer Investigational Site, Skellefteå
  - Pfizer Investigational Site, Stockholm
  - Pfizer Investigational Site, Uddevalla
  - Pfizer Investigational Site, Uppsala
  - Pfizer Investigational Site, Vaxjo
  - Pfizer Investigational Site, Västervik
- United Kingdom (24):
  - Pfizer Investigational Site, Wrexham, Clwyd
  - Pfizer Investigational Site, Woolwich, London
  - Pfizer Investigational Site, Glasgow, Scotland
  - Pfizer Investigational Site, Aberdeen
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Bournemouth
  - Pfizer Investigational Site, Brighton, East Sussex
  - Pfizer Investigational Site, Bristol
  - Pfizer Investigational Site, Cardiff
  - Pfizer Investigational Site, Chichester
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Exeter
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Harrow
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Romford
  - Pfizer Investigational Site, Shrewsbury
  - Pfizer Investigational Site, Warwick

REFERENCES:
- [Derived] Arsenault BJ, Petrides F, Tabet F, Bao W, Hovingh GK, Boekholdt SM, Ramin-Mangata S, Meilhac O, DeMicco D, Rye KA, Waters DD, Kastelein JJP, Barter P, Lambert G. Effect of atorvastatin, cholesterol ester transfer protein inhibition, and diabetes mellitus on circulating proprotein subtilisin kexin type 9 and lipoprotein(a) levels in patients at high cardiovascular risk. J Clin Lipidol. 2018 Jan-Feb;12(1):130-136. doi: 10.1016/j.jacl.2017.10.001. Epub 2017 Oct 12. PMID 29103916
- [Derived] Williams SA, Murthy AC, DeLisle RK, Hyde C, Malarstig A, Ostroff R, Weiss SJ, Segal MR, Ganz P. Improving Assessment of Drug Safety Through Proteomics: Early Detection and Mechanistic Characterization of the Unforeseen Harmful Effects of Torcetrapib. Circulation. 2018 Mar 6;137(10):999-1010. doi: 10.1161/CIRCULATIONAHA.117.028213. Epub 2017 Oct 3. PMID 28974520
- [Derived] Bagdade J, Barter P, Quiroga C, Alaupovic P. Effects of Torcetrapib and Statin Treatment on ApoC-III and Apoprotein-Defined Lipoprotein Subclasses (from the ILLUMINATE Trial). Am J Cardiol. 2017 Jun 1;119(11):1753-1756. doi: 10.1016/j.amjcard.2017.02.049. Epub 2017 Mar 18. PMID 28431663
- [Derived] Barter PJ, Rye KA, Tardif JC, Waters DD, Boekholdt SM, Breazna A, Kastelein JJ. Effect of torcetrapib on glucose, insulin, and hemoglobin A1c in subjects in the Investigation of Lipid Level Management to Understand its Impact in Atherosclerotic Events (ILLUMINATE) trial. Circulation. 2011 Aug 2;124(5):555-62. doi: 10.1161/CIRCULATIONAHA.111.018259. Epub 2011 Jul 18. PMID 21804130
- [Derived] Dogan S, Duivenvoorden R, Grobbee DE, Kastelein JJ, Shear CL, Evans GW, Visseren FL, Bots ML; Radiance 1 and Radiance 2 Study Groups. Ultrasound protocols to measure carotid intima-media thickness in trials; comparison of reproducibility, rate of progression, and effect of intervention in subjects with familial hypercholesterolemia and subjects with mixed dyslipidemia. Ann Med. 2010 Sep;42(6):447-64. doi: 10.3109/07853890.2010.499132. PMID 20645885
- [Derived] Dogan S, Duivenvoorden R, Grobbee DE, Kastelein JJ, Shear CL, Evans GW, Visseren FL, Bots ML; Radiance 1 and 2 Study Groups. Completeness of carotid intima media thickness measurements depends on body composition: the RADIANCE 1 and 2 trials. J Atheroscler Thromb. 2010 May;17(5):526-35. doi: 10.5551/jat.3269. Epub 2010 Mar 13. PMID 20228610
- [Derived] Vergeer M, Bots ML, van Leuven SI, Basart DC, Sijbrands EJ, Evans GW, Grobbee DE, Visseren FL, Stalenhoef AF, Stroes ES, Kastelein JJ. Cholesteryl ester transfer protein inhibitor torcetrapib and off-target toxicity: a pooled analysis of the rating atherosclerotic disease change by imaging with a new CETP inhibitor (RADIANCE) trials. Circulation. 2008 Dec 9;118(24):2515-22. doi: 10.1161/CIRCULATIONAHA.108.772665. Epub 2008 Nov 24. PMID 19029469
- [Derived] Barter PJ, Caulfield M, Eriksson M, Grundy SM, Kastelein JJ, Komajda M, Lopez-Sendon J, Mosca L, Tardif JC, Waters DD, Shear CL, Revkin JH, Buhr KA, Fisher MR, Tall AR, Brewer B; ILLUMINATE Investigators. Effects of torcetrapib in patients at high risk for coronary events. N Engl J Med. 2007 Nov 22;357(21):2109-22. doi: 10.1056/NEJMoa0706628. Epub 2007 Nov 5. PMID 17984165
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5091043&StudyName=A+Study+Examining+Torcetrapib%2FAtorvastatin+And+Atorvastatin+Effects+On+Clinical+CV+Events+In+Patients+With+Heart+Disease